CLINICAL TRIAL: NCT00299533
Title: A Randomized, Double-blind, Placebo-controlled, Prospective Study Evaluating the Usefulness of Polyunsaturated Fatty Acids (PUFA) in Patients Wtih Uncontrolled Epilepsy
Brief Title: Polyunsaturated Fatty Acids for Adjunctive Treatment of Refractory Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: CURE Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-P-000025/14
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Fish Oils

INTERVENTIONS:
Drug: Fish oil (Super Omega-3, 4 caps/d) vs. placebo

SUMMARY:
We are studying whether the addition of fish oil capsules, containing 2.2 gm of polyunsaturated fatty acids, when added to antiepileptic drugs improve seizure control.

DETAILED DESCRIPTION:
Polyunsaturated Fatty Acids for Treatment of Refractory Epilepsy

ABSTRACT

Objective: The primary objective of the study is to determine whether polyunsaturated fatty acids (PUFA) can be used safely and effectively as a treatment for epilepsy.

Background: Patients with intractable epilepsy are often on more than one medication and experience intolerable side effects. Fatty acids have been shown to be protective against seizures in animal models, but there is little human data. Recently, however, a small case series of patients with intractable epilepsy provided evidence of an anti-seizure effect without major side effects. There are no controlled trials of PUFA in humans.

Design/Methods: Patients with uncontrolled partial or generalized epilepsy characterized by at least 4 seizures/month will be randomized to placebo vs. PUFA in a double-blind fashion. Subjects will remain on their current drug(s) while a 4-week baseline seizure count occurs. Dosage will then be titrated over 1 week to 1.1 grams twice daily, and will be followed by a 15-week treatment phase with monthly visits, seizure counts, pill counts, AED levels, adverse event reporting, and neurological examinations. Quality of life will be measured before and after the study using the SF-36 and the QOLIE (Quality of Life in Epilepsy) -31. If subjects wish to continue treatment, they will be given the opportunity at the end of the 20-week period, and those randomized to placebo will have the opportunity to begin treatment with PUFA.

Analysis: The number of subjects achieving a 50% reduction in seizure frequency during the 15-week treatment period relative to the 4-week prospective baseline will be compared for treated vs. control groups using Fisher's exact test. Secondary endpoints will include percent seizure reduction, which will be analyzed using the Mann-Whitney test, and quality of life data, as measured by the SF-36 and QOLIE 31.

Conclusion: There is sufficient preliminary data to suggest that PUFA can be an effective and well-tolerated treatment for epilepsy. If efficacy, safety, and tolerability of PUFA are confirmed, the proposed study will provide the foundation for a larger multi-center trial.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects must have at least one seizure or seizure cluster per week, or at least four per month. They may have partial or generalized epilepsy as diagnosed by a board certified neurologist with subspecialty training in epilepsy. Subjects must be at least 18 years of age, and able to give signed informed consent.

Exclusion Criteria:

* Potential subjects will be considered ineligible for the study if they exhibit frequent vomiting, inability to swallow, an allergy to fatty acids, or a medical condition that could interfere with oral medication intake. Subjects with markedly elevated cholesterol levels (>260) or who receive drugs that affect lipid metabolism, such as HMG CoA inhibitors, will be excluded as well. Due to the theoretical possibility of platelet dysfunction, subjects taking Coumadin® or high doses of aspirin (>325mg daily) will not be considered eligible for the study. Subjects who are pregnant or nursing will also be excluded due to any possible teratogenic effects on the fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-02; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
% of subjects with 50% decrease in seizure frequency

SECONDARY OUTCOMES:
% seizure reduction

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Bromfield, M.D., Principal Investigator — Brigham and Women's Hospital